CLINICAL TRIAL: NCT06313138
Title: Effectiveness of the Individual and Family Health Literacy Enhancement Program Among Older Persons With Physical Multimorbidity
Brief Title: Effectiveness of Health Literacy Enhancement Program Among Older Persons With Physical Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantong University (Other)
Collaborators: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Jun Shan, Phd Candidate, Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NantongJS
Record Dates: First submitted 2024-01-13; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-01

CONDITIONS: Multiple Chronic Conditions；Diabetes；Hypertension
Keywords: Aged; multimorbidity; Health literacy; Self-management.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The Individual and Family Enhancement Program Session 1(1st week): Assessment and exchange information and building trusting relationship between researcher and participants; Session 2-3(1st-2nd week): Information sharing based on PITS model (Pathophysiology, Symptoms, or signs) and evaluation participants' understanding based on UPP scale.
  Session 4-5(2nd-3rd week): Information sharing based on PITS model (treatment) and health maintenance skills.
  Session 6 (3rd week): Information sharing based on PITS model (specifics) and family role in self-management.
  Session7(4th week): Evaluation and summary. Session 8(5th week): Assess health literacy and information provision
  Interventions: Other: The Individual and Family Enhancement Program
- control group (Other): Community nurses provide usual care
  Interventions: Other: The Individual and Family Enhancement Program

INTERVENTIONS:
Other: The Individual and Family Enhancement Program — The program is a group-based intervention which will be developed by the researcher based on the Individual and Family Self-Management Theory (IFSMT) (self-management skills) and the principle of Medagogy (PITS model: Pathophysiology, Indications, Treatments, Specifies) to improve patients' and their families' understanding of disease-related information and self-management skills consisting of goal setting and action plan, self-monitoring, solving problems and decision-making, and emotional control.

SUMMARY:
The study aims to examine the effectiveness of individual and family health literacy enhancement program among older persons with physical multimorbidity.

Specific objectives are:

1. To compare self-management, treatment burden, and symptom burden of older persons with physical multimorbidity between before and after receiving the individual and family health literacy enhancement program.
2. To compare self-management, treatment burden, and symptom burden of older persons with physical multimorbidity between those receiving the individual and family health literacy enhancement program and those receiving usual care.

Participants in the control group will receive usual care by physician and nurses during the experimental period. The usual care consists of physical examination, regular treatment protocol, patient education and telephone follow-up by community nurses.

Participants in the interventional group will receive the program which is a group-based intervention developed by the researcher based on the Individual and Family Self-Management Theory (IFSMT) (self-management skills) and the principle of Medagogy (PITS model: Pathophysiology, Indications, Treatments, Specifies) to improve patients' and their families' understanding of disease-related information and self-management skills consisting of goal setting and action plan, self-monitoring, solving problems and decision-making, and emotional control.The program will be divided into 8 sessions. Each session will be lasted for 2 hours with 1 intermittent break (10 minutes), and it will be held twice a week, and the last session will be held 1 week after the 7th session. Therefore, it will last for 5 weeks in total.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years old;
* Having been diagnosed with hypertension and type 2 diabetes for at least 6 months;
* Being able to read and write Chinese language;
* Cognitive intact as measured by the Mini-Mental State Examination (MMSE) with the score ≥ 24;
* Physically independence as measured by the Barthel ADL Index and the score above 12 out of 20 ;
* Willing to participate in the study;
* Having at least a family member who is willing to participate in the study.

Exclusion Criteria:

* Having other diseases or severe complications from their health problems that making them unable to fully participate through all process of the program including ischemic heart disease, myocardial infarction, heart failure, stroke, acute renal failure, diabetic ketoacidosis, and diabetic coma;

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Self-management | 8 weeks after intervention completion
  Self-management will be measured by Partners in Health (PIH) Scale for older persons with physical multimorbidity which was originally developed by Battersby et al in 2003 and translated into Chinese by Chiu in 2017. The possible total score was between 0 and 96. A higher total score indicates patients with better self-management knowledge and behaviors.
Treatment burden | 12 weeks after intervention completion
  Treatment burden will be measured by the Treatment Burden Questionnaire (TBQ) initially developed and validated in the France by Tran (2012) and translated into Chinese by Zhang (2021). Each item is scored from 0(not problem) to 10 (big problem) with total scores ranging from 0 (no burden) to 150(high burden). A higher score indicates higher treatment burden.
Symptom burden | 12 weeks after intervention completion
  Symptom burden will be measured by The Memorial Symptom Assessment Scale Short Form MSAS(MSAS-SF) initially developed by Chang et al (2000) and translated into simplified Chinese language by Fu et al (2018). The total score is the average severity of symptoms within past week, with symptoms not experienced scored as a zero. A higher score equates to greater symptom burden.

SECONDARY OUTCOMES:
Health literacy | 1 week after intervention completion
  Health literacy will be measured by the functional Communication Critical Health Literacy (FCCHL) for older persons with physical multimorbidity which was originally developed by Ishikawa et al (2008) and translated into Chinese by Zhao XY(2021). The total health literacy scale wasformed by adding all fourteen items. Each item is rated on a 4-point Likert scale, ranging from 1 (never) to 4 (often), with a higher score reflecting abundant health literacy.
  be used to monitor the intermediate outcome of the program implementation and will be measured by the functional Communication Critical Health Literacy (FCCHL)(Ishikawa, Takeuchi, & Yano, 2008) for older persons with physical multimorbidity which was originally developed by Ishikawa et al (2008) and translated into Chinese by Zhao XY(2021)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shan, Principal Investigator — Nantong University
Locations (1):
- Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT06313138/ICF_000.pdf